CLINICAL TRIAL: NCT01969097
Title: Efficacy Basics of Bihemispheric Motorcortex Stimulation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MotorCtx-Stroke-tDCS
Record Dates: First submitted 2013-10-07; First posted 2013-10-25 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Stroke; Hemiparesis
Keywords: Stroke; Hemiparesis; tDCS; Motor cortex
MeSH Terms: conditions — Stroke; Paresis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dual tDCS + motor training (Experimental): Motor training of the affected upper extremity combined with dual transcranial direct current stimulation (tDCS).
  Interventions: Device: tDCS; Behavioral: Motor training
- Anodal tDCS + motor training (Active Comparator): Motor training of the affected upper extremity combined with anodal tDCS.
  Interventions: Device: tDCS; Behavioral: Motor training
- Sham tDCS + motor training (Sham Comparator): Motor training of the affected upper extremity combined with sham tDCS.
  Interventions: Device: tDCS; Behavioral: Motor training

INTERVENTIONS:
Device: tDCS — transcranial direct current stimulation (tDCS)
Behavioral: Motor training — Motor training of the affected upper extremity (5 days, 25 min/day).

SUMMARY:
The aim of the study is to investigate whether the combination of bihemispheric ("dual") transcranial direct current stimulation (tDCS) and motor training on 5 consecutive days facilitates motor recovery in chronic stroke. Results will be compared to a matched group of patients undergoing anodal tDCS as well as a control group receiving sham tDCS. Functional and structural magnetic resonance imaging (MRI) before/after the intervention and during a 3 month follow-up will help investigating neural correlates of expected changes in motor function of the affected upper extremity.

ELIGIBILITY:
Inclusion Criteria:

* chronic stroke (>6 months after stroke)
* age: 18 to 80 years
* non-hemorrhagic or hemorrhagic stroke

Exclusion Criteria:

* more than 1 stroke
* severe alcohol disease or drug abuse, severe psychiatric disease like depression or psychosis
* severe cognitive deficits
* severe untreated medical conditions
* other neurologic diseases
* severe microangiopathy
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Motor Function of the Affected Upper Extremity | Change from baseline after 5 days (immediately after intervention)
  Effects of dual tDCS + training vs sham-tDCS + training on the motor function of the affected upper extremity (measured by standardized behavioral tests).
Motor Function of the Affected Upper Extremity | change from baseline after 3 months
  Effects of dual tDCS + training vs sham-tDCS + training on the motor function of the affected upper extremity (measured by standardized behavioral tests).

SECONDARY OUTCOMES:
Motor Function of the Affected Upper Extremity | After 5 days (immediately after intervention), after 3 months vs baseline (before intervention)
  Effects of dual tDCS + training vs anodal tDCS + training on the motor function of the affected upper extremity (measured by standardized behavioral tests).
Functional Magnetic Resonance Imaging | After 5 days (immediately after intervention), after 3 months vs baseline (before intervention)
  Effects of dual tDCS + training vs anodal tDCS + training vs sham-tDCS + training on task-specific activations and functional connectivity (measured by functional Magnetic Resonance Imaging, fMRI).
Diffusion Tensor Imaging | After 5 days (immediately after intervention), after 3 months vs baseline (before intervention)
  Effects of dual tDCS + training vs anodal tDCS + training vs sham-tDCS + training on cerebral microstructure (measured by Diffusion Tensor Imaging, DTI).
Transcranial Magnetic Stimulation | After 5 days vs baseline (before intervention)
  Effects of dual tDCS + training vs anodal tDCS + training vs sham tDCS + training on excitability of the primary motor cortex (measured by Motor Evoked Potentials, MEP, using Transcranial Magnetic Stimulation, TMS).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lindenberg, M.D., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Lindenberg R, Renga V, Zhu LL, Nair D, Schlaug G. Bihemispheric brain stimulation facilitates motor recovery in chronic stroke patients. Neurology. 2010 Dec 14;75(24):2176-84. doi: 10.1212/WNL.0b013e318202013a. Epub 2010 Nov 10. PMID 21068427
- [Background] Lindenberg R, Nachtigall L, Meinzer M, Sieg MM, Floel A. Differential effects of dual and unihemispheric motor cortex stimulation in older adults. J Neurosci. 2013 May 22;33(21):9176-83. doi: 10.1523/JNEUROSCI.0055-13.2013. PMID 23699528
- [Background] Floel A. tDCS-enhanced motor and cognitive function in neurological diseases. Neuroimage. 2014 Jan 15;85 Pt 3:934-47. doi: 10.1016/j.neuroimage.2013.05.098. Epub 2013 May 30. PMID 23727025
- [Derived] Taud B, Lindenberg R, Darkow R, Wevers J, Hofflin D, Grittner U, Meinzer M, Floel A. Limited Add-On Effects of Unilateral and Bilateral Transcranial Direct Current Stimulation on Visuo-Motor Grip Force Tracking Task Training Outcome in Chronic Stroke. A Randomized Controlled Trial. Front Neurol. 2021 Nov 11;12:736075. doi: 10.3389/fneur.2021.736075. eCollection 2021. PMID 34858310
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411